CLINICAL TRIAL: NCT01885637
Title: DOMUS: A Randomized Controlled Clinical Trial of Accelerated Transition From Oncological Treatment to Continuing Palliative Care at Home
Brief Title: DOMUS: A Trial of Accelerated Transition From Oncological Treatment to Continuing Palliative Care at Home
Acronym: DOMUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other); TRYG Foundation (Other); The Danish Institute for Health Services Research, Copenhagen, Denmark (Unknown); University of Copenhagen (Other); Danish Knowledge Centre for Palliative Care, Copenhagen, Denmark (Unknown)
Responsible Party: Principal Investigator, Per Sjogren, Professor, M.D., Dr. Med. Sci, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-4-2013-016; 2007--58--0015 (Other: The Danish Data Protection Agency)
Record Dates: First submitted 2013-06-17; First posted 2013-06-25 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Incurable Cancer
Keywords: Palliative; Palliation; Cancer; Care; SPC; Caregivers; Home Care Services, Hospital-Based; Psychological; From Oncological Treatment to Palliative Care at Home; Place of death
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): In the control group, the patients continue to be attached to the health care system in line with current practice. This means that the patient typically remains in hospital or ambulatory and may have contact with one or more hospitals, GP and possibly homecare later in the process. Caregivers in the control group may receive psychological counseling through referral from a GP.
- Intervention Group (Other): Accelerated transition program from oncological treatment to continuous specialized palliative care and psychological intervention at home for incurable cancer patients
  Interventions: Other: Transition program

INTERVENTIONS:
Other: Transition program — Accelerated transition program from oncological treatment to continuous specialized palliative care and psychological intervention at home for incurable cancer patients
  Arms: Intervention Group

SUMMARY:
Danish studies have shown that the majority of palliative cancer patients wish to be cared for and spend the rest of their lives at home. Nevertheless > 50% of palliative cancer patients die in acute hospitals and these figures are found in countries with a highly developed palliative care service as well. Some studies have suggested that, among other causes, delays in the discharge process represent a significant obstacle for achieving care and treatment, and ultimately death at home. Therefore, this randomized controlled trial (RCT) aims at investigating an accelerated transition program from oncological treatment to continuous specialized palliative care at home for patients with incurable cancer. The primary objective of the study is to investigate whether an accelerated transition from oncology care to palliative home care significantly increases home care and death. The secondary objectives are to investigate whether the intervention improves symptom control and quality of life, increases survival, affects health care expenses, improves caregiver quality of life and burden, dyadic coping and grief outcomes. The study will take place in the departments of oncology at Rigshospitalet, where palliative cancer patients will enter the intervention or usual care arms. The intervention is an accelerated transition program, which consists of planning palliative home care and if needed optimization of facilities at home, and a transfer to home care within 5 days of informed consent. On day 1 at home the patient, informal caregiver, nurse, representatives of the specialized palliative care team and if possible the general practitioner and project psychologist meet to organize home care. A dyadic psychological intervention is offered to patients and their informal caregiver during specialized palliative care at home and to bereaved caregivers. The control group will be treated according to the usual principles, but if inadequate palliative care is observed in this group, the study group is obliged to involve responsible professionals. Both groups will be followed by assessments of the patient and the caregiver for up to 6 months and the caregivers 19 month after the patient's death.

DETAILED DESCRIPTION:
The trial is a controlled, randomized clinical trial in which 340 in- and outpatients in the Department of Oncology, at Rigshospitalet (Copenhagen University Hospital), are randomly assigned to either an accelerated transition process from oncological treatment to continuing specialised palliative care (SPC) at home plus standard care or standard care alone.

Patients are randomized immediately after their consent and will be discharged within a maximum of 5 working days from randomization. If these timelines are exceeded due to practical issues, the patient can participate in the trial if he/she completes a new base-line questionnaire (Quality of life questionnaire - Core (EORTC-QLQ-C30), Edmonton Symptom Assessment System (revised version) (ESAS-r), Hospital Anxiety and Depression Scale (HADS), Symptoms priority list, Symptom Checklist-92 (SCL-92), Medical Outcomes Study Social Support Survey (mMOS-SS), Dyadic Coping Inventory (DCI)and Relationship ladder, and still meets the inclusion criteria.

Data collection from patients and informal caregivers:

Patients are identified, informed about the study and consenting patients and their informal caregivers complete questionnaires (baseline), after which patients are randomized to either the intervention or the control group. The intervention group will be assigned a specialised palliative care team (SPT) no later than 5 days after randomization. The control group will continue their current treatment. Two weeks after baseline, patients and caregivers complete questionnaires for the 2-week follow-up. Likewise, the follow-up at 4 and 8-weeks consists of questionnaires completed by patients and caregivers. Six months after baseline, the patient's vital status is retrieved. If the patient is still alive questionnaires are sent to the patient and caregiver.

In case of admissions of the patients in both groups, data regarding causes of admission are retrieved from medical records.

Throughout the psychological intervention, the psychologists will register the thematic content of the sessions.

Data collection from informal caregivers includes the Medical Outcomes Study SF-36, Symptom Checklist-92 (SCL-92), modified Medical Outcomes Study Social Support Survey (mMOS-SSS), Zarit Burden Interview (ZBI), Dyadic Coping Inventory (DCI), Relationship Ladder, and Experiences in Close Relationships-Short Form (ECR-S). Data collection from caregivers will continue after the patient's death in the form of questionnaires, which are to be completed after 14 days, 2, 7, 13 and 19 months into the bereavement process (Medical Outcomes Study SF-36, Symptom Checklist-92 (SCL-92),Pittsburgh Sleep Quality index (PSQI), modified Medical Outcomes Study Social Support Survey (mMOS-SSS), Inventory of Daily Widowed Life (IDWL), Experiences in Close Relationships-Short Form and Prolonged Grief(PG-13)). Further, data on caregivers' use of healthcare services will be retrieved from the National Health Care Register, National Patient Registry, the Psychiatric Central Register and Medicinal Product Statistics Register. After the last session, short semi-structured interviews will be conducted among a selected group of caregivers to identify the elements of the intervention that were experienced as helpful, and to investigate the caregivers' experience of having cared for their relatives at home and their bereavement process.

Blood samples from a subgroup of caregivers:

To analyze Telomere length, 10-milliliter (ml) blood samples from caregivers will be collected in a heparinized glass before and after the intervention. The white blood cells (leukocytes) are isolated and frozen to - 80 degrees Celsius. Blood samples are taken before randomization and after termination of the intervention. When the investigation is complete and all blood samples have been obtained and frozen, we will follow a standard protocol for isolation of telomere DNA. This protocol describes how DNA is analyzed for TL in the leukocytes by using a quantitative polymerase chain reaction (PCR), and how the total average TL is calculated from both the amount of telomeric product, and each copy gene.

The intervention:

1. Before the patient agrees to participate, an information meeting will be held. If the patient gives consent to participate, the CRFs will be completed, the blood sample taken from the caregiver and the patient will be randomized.
2. At day one or two after randomization the research nurse, the patient and informal caregiver discuss the patient's wishes for specialised palliative care in their own home and how these can be reconciled with the caregiver's wishes. The patient and caregiver's perceptions of challenges and concerns related to home care are explored and addressed.
3. Immediately after the planning meeting the conditions in the home are optimized, if needed.
4. Four to five days after randomization a home conference is held with the patient and caregiver, representatives of the SPT, nurse, and as far as possible with the patient's GP and the project psychologist. The SPT in collaboration with the GP and district nursing is now responsible for the distribution of tasks related to treatment and care.
5. Patient and caregiver (the primary informal caregiver, appointed by the patient), will be offered a psychological intervention as part of the multi-disciplinary intervention. The psychological intervention will be guided by an intervention manual developed specifically for the study. After the patient's death, bereaved caregivers will be offered one or two additional session, concluding the intervention.

Elements of the psychological intervention:

The psychological intervention will provide a continuum of sessions both before and after the patient's death, so caregivers continue to be supported after the death of their loved ones. The session content will depend on the specific situation and needs of each patient-caregiver dyad. The sessions may thus address several themes that can support the patient in being at home, for example, communication between the patient and the caregiver, reconciliation of different expectations and wishes for being cared for at home, psycho-education about stress and coping and focus on caregivers' self-care. The psychologist may also serve as a navigator in the event of unresolved issues and problems (i.e. help patients and caregivers to identify the most important issues for them and the right people to contact).

The duration of the study:

The study is completed when 340 patients have been randomized into the study and after the last patient has been followed six months after baseline. Patients in the intervention group can then choose to continue with the SPT after the study completion.

Duration of the study of caregivers ranges from randomization to the end of follow-up 19 months after the death of the patient.

In the control group, the patients continue to be attached to the health care system in line with current practice. This means that the patient typically remains in hospital or ambulatory clinic and may have contact with one or more hospitals, GP and possibly homecare later in the process. Caregivers in the control group may receive psychological counseling through referral from a GP.

ELIGIBILITY:
Inclusion Criteria:

* Adult (at least 18 year old) cancer patients connected to the Department of Oncology, Copenhagen University Hospital
* Patients who want to spend as much time as possible in their own homes supported by an SPT
* Patients with incurable cancer
* Patients with no or limited antineoplastic treatment options or patients who resign antineoplastic treatment
* Patients living in the Capital Region
* Written informed consent

Exclusion Criteria:

* Patients who have already been referred to an SPT
* Hospitalized patients who are not judged capable of being discharged home
* Patients who are admitted to other hospitals
* Patients who do not speak Danish well enough to answer the questionnaires
* Patients who are considered incapable of cooperating in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2013-06; Primary Completion 2017-02 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Place of care and death | Up to 4.5 years
  To investigate whether the transition process and SPC at home in patients with incurable cancer results in more patients in accordance with his/her own request obtains treatment, care, and death in their own homes.

SECONDARY OUTCOMES:
HRQL | Up to 4.5 years
  Whether there is a difference between intervention - and the control groups in change from baseline to the weighted average of 2, 4 and 8-week follow up ("mixed-effect" regressions model) for symptoms / problems and quality of life measured with EORTC QLQ-C30 and The Edmonton Symptom Assessment System (ESAS) and for anxiety and depression measured by HADS. In addition, patients will be asked to prioritize their symptoms after how annoying they are according to a list of symptoms / side effects.
Use of medicine | Up to 4.5 years
  Whether there is a difference between the intervention and control groups in the change from baseline to the weighted average of 2, 4 and 8-week follow up ("mixed-effect" regressions model) in medication use.
Survival time | Up to 4.5 years
  Whether there are differences in the proportion surviving in the two groups and whether the survival time is different between the 2 groups.
Healthcare services and informal care | Up to 4.5 years
  Whether there are differences in resource use (healthcare services and informal care) between the two groups.
Cooperation and quality of the process | Up to 4.5 years
  Whether there is a difference between the professionals' assessments of cooperation and quality of the process in the intervention and control groups.
Anxiety and depression | Up to 4.5 years
  Whether patients in the intervention group will have less anxiety and depression than patients in the control group.
Caregiver: anxiety and depression | Up to 4.5 years
  Whether there is a difference between caregivers in the intervention and control groups in the change from baseline to 2, 4 and 8-week follow up in anxiety and depression (as assessed by the SCL-92), and whether there is a difference in anxiety and depression between caregivers in the intervention and control groups at follow-up 2 weeks, 2, 7, 13, and 19 months after bereavement.
Caregiver: prolonged grief | Up to 4.5 years
  Whether caregivers in the intervention group will less frequently exhibit prolonged grief (as measured by the PG-13 questionnaire) and have fewer symptoms of prolonged grief than caregivers in the control group at follow-up assessments at 2 weeks, 2, 7, 13, and 19 months after bereavement.
Dyadic coping | Up to 4.5 years
  Whether there is a difference between patient and caregiver dyads in the intervention and control groups in the change from baseline to 2, 4 and 8-week follow up in dyadic coping (as assessed by subscales of the Dyadic Coping Inventory (DCI)).
Preference for place of treatment and care | Up to 4.5 years
  Whether there will be a difference in the preference for place of treatment and care between patients and caregivers in the intervention and control groups, as assessed at baseline and the 2, 4, and 8 week follow-up.
Caregiver: HRQoL | Up to 4.5 years
  Whether there is a difference between caregivers in the intervention and control group in the change from baseline to 2, 4 and 8-week follow up in health related quality of life, as measured by the SF-36 (incl. subscales) , and between bereaved caregivers in the intervention and control group at 2 weeks, 2, 7, 13, and 19 months after bereavement.
Caregiver: Use of health services | Up to 4.5 years
  Whether there is a difference in use of health care services between caregivers in the intervention and control group, as obtained from registers.
Caregiver burden | Up to 4.5 years
  Whether there is a difference between caregivers in the intervention and control groups in the change from baseline to 2, 4 and 8-week follow up in caregiver burden, as measured by the Zarit Burden Interview (ZBI).
Caregiver: telomere degradation | Up to 4.5 years
  Whether telomere degradation will be lower and telomerase activity higher between baseline and 2 months after bereavement among caregivers in the intervention group than among caregivers in the control group.
Caregiver: The psychological intervention | Up to 4.5 years
  Within the intervention group, it will be examined which elements of the psychological intervention were experienced as meaningful / efficacious by the bereaved caregivers after the intervention.
Caregiver Grief | Up to 4.5 years
  Whether there will be a difference in bereaved caregivers' grief in the intervention and control group, as measured by the Inventory of Daily Widowed Life(IDWL) (and its subscales) at 2 weeks, 2, 7, 13, and 19 months after bereavement.
Caregiver health behavior | Up to 4.5 years
  Whether there is a difference between bereaved caregivers' health behavior in the intervention and control group, as measured by items on alcohol consumption, smoking, meals, and physical activity, and the PSQI at 2 weeks, 2, 7, 13, and 19 months after bereavement.
Hospital admissions | Up to 4.5 years
  Whether there is a difference in cause, number, type, length and outcome of admissions between the groups.
Non-participation | up to 4.5 years
  To investigate differences between participants and non-participants on demographic and clinical characteristics, and self-reported symptom burden, as well as reasons for non-participation in the DOMUS study and their relation to non-participant-characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Per Sjøgren, Proff., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Depatment of Oncology, Rigshospitalet, Copenhagen Ø, Denmark

REFERENCES:
- [Derived] Halling CMB, Wolf RT, Sjogren P, Von Der Maase H, Timm H, Johansen C, Kjellberg J. Cost-effectiveness analysis of systematic fast-track transition from oncological treatment to specialised palliative care at home for patients and their caregivers: the DOMUS trial. BMC Palliat Care. 2020 Sep 15;19(1):142. doi: 10.1186/s12904-020-00645-7. PMID 32933489
- [Derived] Benthien K, Diasso P, von Heymann A, Nordly M, Kurita G, Timm H, Johansen C, Kjellberg J, von der Maase H, Sjogren P. Oncology to specialised palliative home care systematic transition: the Domus randomised trial. BMJ Support Palliat Care. 2020 Sep;10(3):350-357. doi: 10.1136/bmjspcare-2020-002325. Epub 2020 Jul 17. PMID 32680894
- [Derived] von Heymann-Horan A, Bidstrup P, Guldin MB, Sjogren P, Andersen EAW, von der Maase H, Kjellberg J, Timm H, Johansen C. Effect of home-based specialised palliative care and dyadic psychological intervention on caregiver anxiety and depression: a randomised controlled trial. Br J Cancer. 2018 Nov;119(11):1307-1315. doi: 10.1038/s41416-018-0193-8. Epub 2018 Nov 14. PMID 30425351
- [Derived] Nordly M, Skov Benthien K, Vadstrup ES, Kurita GP, von Heymann-Horan AB, von der Maase H, Johansen C, Timm H, Kjellberg J, Sjogren P. Systematic fast-track transition from oncological treatment to dyadic specialized palliative home care: DOMUS - a randomized clinical trial. Palliat Med. 2019 Feb;33(2):135-149. doi: 10.1177/0269216318811269. Epub 2018 Nov 12. No abstract available. PMID 30415608
- [Derived] von Heymann-Horan A, Bidstrup PE, Johansen C, Rottmann N, Andersen EAW, Sjogren P, von der Maase H, Timm H, Kjellberg J, Guldin MB. Dyadic coping in specialized palliative care intervention for patients with advanced cancer and their caregivers: Effects and mediation in a randomized controlled trial. Psychooncology. 2019 Feb;28(2):264-270. doi: 10.1002/pon.4932. Epub 2018 Nov 15. PMID 30353600
- [Derived] Skov Benthien K, Nordly M, von Heymann-Horan A, Rosengaard Holmenlund K, Timm H, Kurita GP, Johansen C, Kjellberg J, von der Maase H, Sjogren P. Causes of Hospital Admissions in Domus: A Randomized Controlled Trial of Specialized Palliative Cancer Care at Home. J Pain Symptom Manage. 2018 Mar;55(3):728-736. doi: 10.1016/j.jpainsymman.2017.10.007. Epub 2017 Oct 19. PMID 29056562
- [Derived] Benthien KS, Nordly M, Videbaek K, Kurita GP, von der Maase H, Timm H, Simonsen MK, Johansen C, Sjogren P. Classification of a palliative care population in a comprehensive cancer centre. Support Care Cancer. 2016 Apr;24(4):1865-73. doi: 10.1007/s00520-015-2979-z. Epub 2015 Oct 13. PMID 26463644
- [Derived] Nordly M, Benthien KS, Von Der Maase H, Johansen C, Kruse M, Timm H, Vadstrup ES, Kurita GP, von Heymann-Horan AB, Sjogren P. The DOMUS study protocol: a randomized clinical trial of accelerated transition from oncological treatment to specialized palliative care at home. BMC Palliat Care. 2014 Sep 9;13:44. doi: 10.1186/1472-684X-13-44. eCollection 2014. PMID 25242890